CLINICAL TRIAL: NCT04460664
Title: Exploratory Assessment of the Coagulation Changes Associated With Severe Inflammation in COVID-19 Patients
Brief Title: Coagulation Changes Associated With COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-035
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: COVID; Disseminated Intravascular Coagulation; Coagulation Disorder
Keywords: Viscoelastic testing; Quantra; COVID-19
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Hemostatic Disorders; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Subjects admitted to floor: COVID-19 patients admitted to the floor as initial place of hospitalization
  Interventions: Diagnostic Test: Quantra System
- Subjects admitted or transferred to ICU: COVID-19 patients admitted to the ICU as initial place of hospitalization or transferred to ICU from floor
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: QPlus Cartridge

SUMMARY:
This study will study the potential utility of the Quantra QPlus System in patients inflicted with COVID-19 disease.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QPlus Cartridge can measure hypocoagulable and hypercoagulable conditions resulting from the functional interaction of the enzymatic and cellular components of coagulation and therefore, can be invaluable for longitudinal monitoring of the coagulopathies reported in COVID-19 patients and the response to anticoagulants.

This single-center, prospective, observational pilot study will characterize changes in the coagulation status of patients with COVID-19 infection during their hospital stay using the Quantra QPlus System.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject has a diagnosis of COVID-19 and has been admitted to the hospital
* Subject has one or more risk factors for a poor outcome with COVID-10 disease: advanced age (>=60 years), morbid obesity, diabetes, COPD, CAD
* Subject, or subject's legally authorized representative is willing and agrees to provide informed consent.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is pregnant
* Subject is incarcerated.
* Subject, or subject's legally authorized representative is unable or unwilling to provide informed consent.
* Subject is affected by a condition that, in the opinion of the treatment team, may pose additional risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be adult (>=18 years) patients with a diagnosis of COVID-19 disease admitted to the hospital for treatment of their disease. Subjects will be enrolled at a ratio of 1 admitted to floor for every 2 admitted to ICU as initial place of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Quantra Clot Time results | Within 24 hours of admission to the hospital
  Coagulation function assessed by the Quantra
Quantra Clot Time results | 48 to 72 hours after transfer to ICU
  Coagulation function assessed by the Quantra
Quantra Clot Time results | 1 to 24 hours prior to discharge from hospital
  Coagulation function assessed by the Quantra
Quantra Clot Stiffness results | Upon arrival at hospital
  Coagulation function assessed by the Quantra
Quantra Clot Stiffness results | 48 to 72 hours after transfer to ICU
  Coagulation function assessed by the Quantra
Quantra Clot Stiffness results | 1 to 24 hours prior to discharge from hospital
  Coagulation function assessed by the Quantra

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No